CLINICAL TRIAL: NCT01725113
Title: A Randomized, Prospective, Cross-Over Study of Calcitriol vs. Paricalcitol in the Treatment of Mineral and Bone Disease in Hemodialysis Patients
Brief Title: Management of Mineral and Bone Disease in Hemodialysis-Calcitriol vs. Paricalcitol
Acronym: ECRIP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Nationwide shortage of study meds in 2013 loss of funding & competing studies
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12027
Record Dates: First submitted 2012-11-07; First posted 2012-11-12 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Kidney Failure; Secondary Hyperparathyroidism; Hyperphosphatemia; Hypercalcemia
MeSH Terms: conditions — Renal Insufficiency; Hyperparathyroidism, Secondary; Hyperphosphatemia; Hypercalcemia | interventions — Calcitriol; paricalcitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcitriol, then Paricalcitol (Experimental): Patients randomized to an active vitamin D treatment protocol based on IV calcitriol. After 14 weeks, patients cross-over to an active vitamin D protocol based on IV paricalcitol for 14 weeks.
  Interventions: Drug: Calcitriol; Drug: Paricalcitol
- Paricalcitol, then Calcitriol (Active Comparator): Patients randomized to an active vitamin D treatment protocol based on IV paricalcitol. After 14 weeks, patients cross-over to an active vitamin D protocol based on IV calcitriol for 14 weeks.
  Interventions: Drug: Calcitriol; Drug: Paricalcitol

INTERVENTIONS:
Drug: Calcitriol — 3 times weekly
  Other Names: Calcijex®
Drug: Paricalcitol — 3 times weekly
  Other Names: Zemplar®

SUMMARY:
The purpose of this non-inferiority study is to compare the safety and effectiveness of a mineral and bone disease treatment protocol based on calcitriol to one based on paricalcitol in hemodialysis patients using revised Kidney Disease: Improving Global Outcomes (KDIGO) parathyroid hormone targets.

DETAILED DESCRIPTION:
Active vitamin D analogs have been the mainstay of treatment for patients on hemodialysis with mineral and bone disease (MBD) for the past decade. Intravenous calcitriol is an active vitamin D analog which is nearly identical to natural 1, 25 Vitamin D3. Calcitriol results from the hydroxylation of previtamin D3 in the liver and kidney. Paricalcitol, 19-nor-1 , 25-dihydroxyvitamin D2, is a newer agent vitamin D analog. This agent is believed to have an effect more specific to the parathyroid gland, and less specific to absorption of calcium and phosphorus from the gut. Although both formulations appear equally effective in suppressing parathyroid hormone (PTH), studies have suggested a greater calcemic effect with intravenous calcitriol as compared to paricalcitol (1). Due to this, paricalcitol is the predominant active vitamin D analog used in hemodialysis patients in the United States. Two recent changes in the management of hemodialysis patients will likely reduce the amount of active vitamin D analogs used in the near future: the liberalization of PTH goals according to international guidelines, (2) and the implementation of bundled payments for dialysis by Medicare. These changes challenge previous studies that have analyzed the safety and efficacy of these medications. The purpose of this prospective, randomized, cross-over study will be to determine whether calcitriol is as safe and effective as paricalcitol in the treatment of MBD in hemodialysis patients using the revised KDIGO parathyroid hormone targets. Our hypothesis is that calcitriol will be as equally safe and effective as paricalcitol in the treatment of MBD in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

- All subjects will have been treated for at least three months on hemodialysis with IV paricalcitol. These subjects must have a most recent calcium level within the normal range, most recent phosphorus level < 8 mg/dL and a most recent PTH between 130-585 pg/mL

Exclusion Criteria:

Patients will be excluded if:

1. age greater than 18
2. active malignancy
3. expected survival greater than 6 months
4. high likelihood of renal transplant during the study period.
5. Low calcium bath
6. prior parathyroidectomy
7. use of calcimimetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shayan Shirazian, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 16 enrolled participants, 3 were removed due to screen failure and 1 patient experienced death before the start of study.
Period: Overall Study
Arm/Group | Calcitriol, Then Paricalcitol | Paricalcitol, Then Calcitriol
Started | 6 | 6
Completed | 5 | 4
Not Completed | 1 | 2
Not completed — Kidney Transplant | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are only available among participants who completed the trial.
Groups:
- Total Participants Who Completed Trial: Participants (n=9) who completed the trial.
Arm/Group | Total Participants Who Completed Trial
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.11 (5.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Calcium Levels at Month 3 Post Calcitriol Treatment Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Calcitriol: Comprises participants who received Calcitriol either in the first 14 weeks or last 14 weeks of the treatment period.
Arm/Group | Calcitriol
Number analyzed (Participants) | 9
mg/dl | 8.78 (0.332)

2. Primary Outcome: Calcium Levels at Month 3 Post Paricalcitol Treatment Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Paricalcitol: Comprises participants who received Paricalcitol either in the first 14 weeks or last 14 weeks of the treatment period.
Arm/Group | Paricalcitol
Number analyzed (Participants) | 9
mg/dl | 8.6 (0.3)

3. Secondary Outcome: PTH Levels at Month 3 Post Calcitriol Treatment Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Calcitriol
Number analyzed (Participants) | 9
pg/dl | 309.58 (183.33)

4. Secondary Outcome: PTH Levels at Month 3 Post Paricalcitol Treatment Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Paricalcitol
Number analyzed (Participants) | 9
pg/dl | 332.83 (146.9)

5. Secondary Outcome: Phosphorus Levels at Month 3 Post Calcitriol Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Calcitriol
Number analyzed (Participants) | 9
mg/dl | 4.09 (0.71)

6. Secondary Outcome: Phosphorus Levels at Month 3 Post Paricalcitol Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Paricalcitol
Number analyzed (Participants) | 9
mg/dl | 4.45 (1.18)

7. Secondary Outcome: Amount of Active Vitamin D Analog Used Through Month 3 Post Calcitriol Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Calcitriol
Number analyzed (Participants) | 9
mcg | 36.9 (34.18)

8. Secondary Outcome: Amount of Active Vitamin D Analog Used Through Month 3 Post Paricalcitol Initiation
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Paricalcitol
Number analyzed (Participants) | 9
mcg | 134.6 (87.35)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Calcitriol | Paricalcitol
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcitriol (N=9) | Paricalcitol (N=9)
Hematuria (Renal and urinary disorders) | 1 | 1 — Hematuira resulting in hospital admission.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes